CLINICAL TRIAL: NCT03264989
Title: A Phase 2, Multicenter, Open-Label Study to Assess PK/PD of SEG101 (Crizanlizumab), With or Without Hydroxyurea/Hydroxycarbamide, in Sickle Cell Patients With Vaso-Occlusive Crisis
Brief Title: Pharmacokinetics and Pharmacodynamics Study of SEG101 (Crizanlizumab) in Sickle Cell Disease (SCD) Patients With Vaso- Occlusive Crisis (VOC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSEG101A2202
Record Dates: First submitted 2017-08-04; First posted 2017-08-29 (Actual); Results first posted 2024-04-23 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: Sickle cell disease; SCD; sickle cell anemia; vaso-occlusive crisis; P-selectin; SEG101; crizanlizumab; monoclonal antibody; Anemia, Sickle Cell; HbS Disease; Hemoglobin SC Disease; Sickle Cell Disorders; Sickling Disorder Due to Hemoglobin S
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Hemoglobin SC Disease | interventions — crizanlizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- crizanlizumab (Experimental): SEG101 (crizanlizumab) drug at a dose of 5.0 mg/kg (or 7.5 mg/kg for exploratory group) by IV infusion.
  Interventions: Drug: crizanlizumab

INTERVENTIONS:
Drug: crizanlizumab — Crizanlizumab was administered IV infusion over 30 minutes at the assigned dose on Week 1 Day 1, Week 3 Day 1, and then Day 1 of every 4-week cycle. Cycle = 28 days
  Other Names: SEG101

SUMMARY:
The purpose of the CSEG101A2202 study was to characterize the Pharmacokinetic (PK) and Pharmacodynamic (PD) of SEG101/crizanlizumab and to evaluate the safety and efficacy of SEG101/crizanlizumab in sickle cell disease (SCD) patients.

DETAILED DESCRIPTION:
Study CSEG101A2202 was designed as a Phase II, multicenter, open-label study. The first 45 patients (to identify 27 evaluable patients) were enrolled to the treatment group crizanlizumab 5.0 mg/kg to complete full Pharmacokinetic/Pharmacodynamic (PK/PD) sampling at week 1 and week 15. In all patients, trough PK/PD samples were collected prior to each dose. In addition, throughout the study (and when possible), all patients had blood drawn for serum to assess PK and PD drawn at times of onset and resolution of each VOC event, fever, or infection. Once the up to 45 patients were enrolled, 12 additional patients were enrolled to the exploratory treatment group and began at 7.5 mg/kg of crizanlizumab.

The study was initiated on 19-Dec-2017. This study provides five years follow up data that fully characterizes the safety, tolerability and treatment effect of the 5.0 mg/kg and 7.5 mg/kg doses of crizanlizumab along with the initially planned PK and PD data.

At the time of study closure, crizanlizumab 5.0 mg/kg was an FDA approved treatment in the United States (US) for patients with sickle-cell disease. Therefore, the patients treated with crizanlizumab 5.0 mg/kg dose were encouraged to transition to commercial supply of crizanlizumab. The patients treated with the not currently approved dose of crizanlizumab 7.5 mg/kg were allowed to join a multi-center, multi-national, rollover clinical trial (Study SEG101A2401B), for continued access to treatment with crizanlizumab.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female patients 16-70 years of age (inclusive)
* Confirmed diagnosis of sickle cell disease by hemoglobin electrophoresis or high-performance liquid chromatography (HPLC) [performed locally]. All sickle cell disease genotypes are eligible.
* Experienced at least 1 VOC within the preceding 12 months prior to Screening, as determined by medical history.
* If receiving HU/HC or erythropoietin stimulating agent, must have been receiving the drug for at least 6 months prior to Screening
* Hemoglobin ≥4.0 g/dL. Absolute neutrophil count ≥1.0 x 109/L and platelet count ≥75 x 109/L
* Adequate renal and hepatic function as defined:
* GFR ≥45 mL/min/1.73 m2 calculated by CKD-EPI
* ALT ≤3 x ULN
* Direct (conjugated) bilirubin ≤2 x ULN
* ECOG performance status ≤2
* Written informed consent (or assent/ parental consent for minor subjects) prior to any screening procedures

Exclusion Criteria:

* History of stem cell transplant.
* Acute VOC ending 7 days prior to first dosing
* Ongoing hospitalization prior to Screening
* Received blood products within 30 days to first dosing
* Participating in a chronic transfusion program (pre-planned series of transfusions for prophylactic purposes)
* History of severe hypersensitivity reactions to other monoclonal antibodies
* Received a monoclonal antibody or immunoglobulin -based agent within 1 year of Screening, or has documented immunogenicity to a prior biologic.
* Received active treatment on another investigational trial within 30 days (or 5 half-lives of that agent, whichever is greater) prior to Screening
* Significant active infection or immune deficiency (including chronic use of immunosuppressive drugs)
* Resting QTcF ≥470 msec at pretreatment (baseline) or other cardiac or cardiac repolarization abnormality

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - Novartis Investigative Site, Orange, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Childrens Healthcare of Atlanta ., Atlanta, Georgia
  - Augusta University Georgia Patient Treatment, Augusta, Georgia
  - University of Maryland Medical Ctr, Baltimore, Maryland
  - Childrens Hospital at Montefiore, The Bronx, New York
  - Duke University Medical Center Patient Treatment, Durham, North Carolina
  - East Carolina University East Carolina University, Greenville, North Carolina
  - Childrens Hospital Of Philadelphia Patient Treatment, Philadelphia, Pennsylvania
  - Medical Uni of South Carolina Medical Univ of SC, Charleston, South Carolina
  - M Francisco Gonzalez MD PA ., Columbia, South Carolina
  - Carolina Blood and Cancer Care of South Carolina, Rock Hill, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kanter J, Mennito S, Nair SM, Manwani D, Kutlar A, Shah N, Keefe D, Madhamshetty H, Nassin M, Reshetnyak E, Mendonza AE, Liles D. Pharmacokinetics, pharmacodynamics, safety, and efficacy of crizanlizumab in patients with sickle cell disease: final results from the phase II SOLACE-adults study. Ther Adv Hematol. 2024 Nov 3;15:20406207241292508. doi: 10.1177/20406207241292508. eCollection 2024. PMID 39497751
- [Derived] Sy SKB, Tanaka C, Grosch K. Population Pharmacokinetics and Pharmacodynamics of Crizanlizumab in Healthy Subjects and Patients with Sickle Cell Disease. Clin Pharmacokinet. 2023 Feb;62(2):249-266. doi: 10.1007/s40262-022-01193-4. Epub 2022 Dec 18. PMID 36529836
- [Derived] Kanter J, Brown RC, Norris C, Nair SM, Kutlar A, Manwani D, Shah N, Tanaka C, Bodla S, Sanchez-Olle G, Albers U, Liles D. Pharmacokinetics, pharmacodynamics, safety, and efficacy of crizanlizumab in patients with sickle cell disease. Blood Adv. 2023 Mar 28;7(6):943-952. doi: 10.1182/bloodadvances.2022008209. PMID 36355805
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1912

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 patients were enrolled sequentially to study the at 5 mg/kg arm and at 7.5 mg/kg.
Pre-assignment Details: This study was conducted in 12 centers in the United States only.
Groups:
- Crizanlizumab 5.0 mg/kg: Participants were administered crizanlizumab at a dose of 5.0 mg/kg by IV infusion.
- Crizanlizumab 7.5 mg/kg: Participants were administered crizanlizumab at a dose of 7.5 mg/kg by IV infusion.
Period: Overall Study
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg
Started | 45 | 12
Completed (Completed = Treatment ongoing. Not Completed = Discontinued from treatment) | 0 | 0
Not Completed | 45 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — New Therapy for study Indication | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Patient decision | 13 | 0
Not completed — Physician Decision | 6 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Death | 1 | 1
Not completed — Pregnancy | 2 | 0
Not completed — End of Study | 19 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): Consisted of all patients to whom crizanlizumab had been assigned and who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg | Total
Number analyzed (Participants) | 45 | 12 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (12.71) | 26.8 (12.25) | 31.2 (12.71)
Age, Customized [Number; unit: participants]
  16 - < 18 years | 1 | 2 | 3
  18 - < 65 years | 43 | 10 | 53
  65 - < 70 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 6 | 31
  Male | 20 | 6 | 26
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 44 | 12 | 56
  White and Black or African American | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK): AUCd15 and AUCtau of Crizanlizumab at 5.0 mg/kg in Sickle Cell Disease (SCD) Patients
Description: To characterize PK of crizanlizumab at 5.0 mg/kg in SCD patients. AUCd15: The AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1) after single dose AUCtau: The AUC calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1)
Time Frame: 1st dose: Day 1: (pre-dose, 0.5, 1, 2, 4, 6 & 24 hours post dose, Days 4, 8 & 15; 5th dose: Day 1 (pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post dose), Days 4, 8, 15, 22 & 29
Population: The PK analysis set 1 (PAS1) included all patients who provided at least one evaluable PK profile in the 5.0 mg/kg arm.
Measure: Mean (Standard Deviation); unit: hr*μg/mL
Arm/Group | Crizanlizumab 5.0 mg/kg
Number analyzed (Participants) | 45
hr*μg/mL
  Starting dose (Week 1): AUCd15: number analyzed (Participants) | 38
  Starting dose (Week 1): AUCd15 | 13100 (2810)
  Steady State (Week 15): AUCtau: number analyzed (Participants) | 35
  Steady State (Week 15): AUCtau | 20800 (5030)

2. Primary Outcome: PK: Cmax of Crizanlizumab at 5.0 mg/kg in Sickle Cell Disease (SCD) Patients
Description: To characterize PK of crizanlizumab at 5.0 mg/kg in SCD patients. Cmax: The maximum (peak) observed serum drug concentration after dose administration (mass x volume-1).
Time Frame: After the starting dose (Week 1) and after multiple doses (steady state, Week 15)
Population: The PK analysis set 1 (PAS1) included all patients who provided at least one evaluable PK profile in the 5.0 mg/kg arm. The Cmax analysis was done on all participants including those for at starting dose (n =42) and steady state (n = 36).
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Crizanlizumab 5.0 mg/kg
Number analyzed (Participants) | 45
μg/mL
  Starting dose (Week 1): number analyzed (Participants) | 42
  Starting dose (Week 1) | 102 (29.8)
  Steady State (Week 15): number analyzed (Participants) | 36
  Steady State (Week 15) | 123 (36.4)

3. Primary Outcome: Pre-dose Concentrations Prior to Each Study Drug Dose
Description: To characterize PK of crizanlizumab at 5.0 mg/kg in SCD patients, by serum concentrations by treatment group.
  Data was collected prior to each study drug dose; From Week 3 (loading dose), pre-dose (trough) concentrations were obtained every 4 weeks.
Time Frame: Pre-dose at Day 1 on Weeks 3, 7, 11, 15, 19, 23, 27, 31, 35, 39, 43, 47, 51
Population: PK Analysis set 2 (PAS2): Included all patients who received at least one planned treatment of 5 mg/kg and provided at least one corresponding evaluable PK concentration.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Crizanlizumab 5.0 mg/kg
Number analyzed (Participants) | 45
μg/mL
  Week (W) 3 Day 1 (D)1: 0 hrs pre-dose: number analyzed (Participants) | 38
  Week (W) 3 Day 1 (D)1: 0 hrs pre-dose | 18.0 (6.42)
  W7 D1: 0 hrs pre-dose: number analyzed (Participants) | 42
  W7 D1: 0 hrs pre-dose | 10.8 (5.21)
  W11 D1: 0 hrs pre-dose: number analyzed (Participants) | 41
  W11 D1: 0 hrs pre-dose | 9.04 (5.04)
  W15 D1: 0 hrs pre-dose: number analyzed (Participants) | 38
  W15 D1: 0 hrs pre-dose | 10.0 (5.39)
  W19 D1: 0 hrs pre-dose: number analyzed (Participants) | 36
  W19 D1: 0 hrs pre-dose | 9.37 (4.95)
  W23 D1: 0 hrs pre-dose: number analyzed (Participants) | 41
  W23 D1: 0 hrs pre-dose | 9.91 (5.09)
  W27 D1: 0 hrs pre-dose: number analyzed (Participants) | 40
  W27 D1: 0 hrs pre-dose | 9.65 (4.03)
  W31 D1: 0 hrs pre-dose: number analyzed (Participants) | 40
  W31 D1: 0 hrs pre-dose | 9.75 (4.66)
  W35 D1: 0 hrs pre-dose: number analyzed (Participants) | 39
  W35 D1: 0 hrs pre-dose | 9.48 (4.60)
  W39 D1: 0 hrs pre-dose: number analyzed (Participants) | 40
  W39 D1: 0 hrs pre-dose | 9.54 (5.47)
  W43 D1: 0 hrs pre-dose: number analyzed (Participants) | 39
  W43 D1: 0 hrs pre-dose | 8.53 (5.24)
  W47 D1: 0 hrs pre-dose: number analyzed (Participants) | 40
  W47 D1: 0 hrs pre-dose | 8.96 (4.31)
  W51 D1: 0 hrs pre-dose: number analyzed (Participants) | 39
  W51 D1: 0 hrs pre-dose | 8.45 (4.88)

4. Primary Outcome: Percentage of P-selectin Inhibition After the Starting Dose (PD-AUCd15), After Multiple Doses (PD-AUCd29) of Crizanlizumab at 5.0 mg/kg in Sickle Cell Disease (SCD) Patients
Description: PD-AUCd15 and PD-AUCd29 were derived from the P-selectin inhibition data of week 1 and week 15, respectively.
  To characterize PD of crizanlizumab at 5.0 mg/kg in SCD patients The area under the curve (AUC) of percentage of P-selectin inhibition versus time profile after the starting dose (PD-AUCd15) and after multiple doses (PD-AUCd29) is being reported.
Time Frame: 1st dose: Day 1: (pre-dose, 0.5, 1, 2, 4, 6 & 24 hours post dose, Days 4, 8, 15; 5th dose: Day 1(pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post dose), Days 4, 8, 15, 22 & 29
Population: PDS1 included all patients who provided at least 1 evaluable PD profile. The P-selectin inhibition analysis was done on all participants including those starting dose (n = 36) and steady state (n = 33).
Measure: Mean (Standard Deviation); unit: hours*% of P-selectin inhibition
Arm/Group | Crizanlizumab 5.0 mg/kg
Number analyzed (Participants) | 43
hours*% of P-selectin inhibition
  Starting dose (Week 1): PD-AUCd15: number analyzed (Participants) | 36
  Starting dose (Week 1): PD-AUCd15 | 33200 (1830)
  Steady state (Week 15): PD-AUCd29: number analyzed (Participants) | 33
  Steady state (Week 15): PD-AUCd29 | 66900 (5540)

5. Secondary Outcome: Annualized Rate of Vaso-occlusive Crisis (VOC) Events Leading to Healthcare Visit in Clinic/Emergency Room (ER)/Hospital
Description: To assess the efficacy of crizanlizumab at 5.0 mg/kg and 7.5 mg/kg in Sickle cell disease (SCD) patients. Annualized rate of VOC=(Number of VOC reported until End date ×365.25)/(End date - date of first dose of study treatment+1).
  End date is defined as the minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-glutamine or other therapies such as voxelotor and erythropoietin to treat SCD and or to prevent/reduce VOCs, cut-off date).
Time Frame: Baseline (Week 1) through approx. 45 months (median exposure to treatment)
Population: The Full analysis set (FAS) consisted of all patients to whom crizanlizumab had been assigned and who received at least one dose of study treatment.
Measure: Median (Full Range); unit: number of events per year
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg
Number analyzed (Participants) | 45 | 12
number of events per year
  Baseline annualized rate of VOC | 4.00 [1.0 to 25.0] | 2.00 [1.0 to 9.0]
  Annualized rate of VOC on treatment | 2.75 [0.0 to 17.3] | 0.97 [0.0 to 7.9]

6. Secondary Outcome: Annualized Rate of VOC Events Treated at Home (Based on Documentation by Health Care Provider Following Phone Contact With Patient)
Description: To assess the efficacy of crizanlizumab at 5.0 mg/kg and 7.5 mg/kg in SCD patients. Annualized rate of VOC=(Number of VOC reported until End date ×365.25)/(End date - date of first dose of study treatment+1).
  End date is defined as the minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-glutamine or other therapies such as voxelotor and erythropoietin to treat SCD and or to prevent/reduce VOCs, cut-off date).
Time Frame: Baseline (Week 1) through approx. 45 months (median exposure to treatment)
Population: The Full analysis set (FAS) consisted of all patients to whom crizanlizumab had been assigned and who received at least one dose of study treatment. The annualized rate of VOC events treated at home analyzed all participants including those who had a VOC event treated at home in the Crizanlizumab 5.0 mg/kg arm and in the Crizanlizumab 7.5 mg/kg arm.
Measure: Median (Full Range); unit: number of events per participant-year
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg
Number analyzed (Participants) | 45 | 12
number of events per participant-year | 0.68 [0.21 to 2.17] | 0.71 [0.35 to 1.74]

7. Secondary Outcome: Annualized Rate of Total and VOC-related Hospitalizations and Emergency Room (ER) Visits
Description: To assess the efficacy of crizanlizumab at 5.0 mg/kg and 7.5 mg/kg in SCD patients. Annualized rate of hospitalizations and ER visits = number of hospitalizations and ER visits reported until end date × 365.25/(End date - treatment start date + 1).
  End date is defined as the minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-glutamine or other therapies such as voxelotor and erythropoietin to treat SCD and or to prevent/reduce VOCs, cut-off date).
Time Frame: Baseine (Week 1) through approx. 45 months (median exposure to treatment)
Population: as for outcome 5
Measure: Median (Full Range); unit: number of events per participant-year
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg
Number analyzed (Participants) | 45 | 12
number of events per participant-year
  Annualized rate (total) | 3.42 [0.0 to 57.8] | 2.47 [0.0 to 8.1]
  Annualized rate (VOC related) | 3.34 [0.0 to 57.8] | 0.86 [0.0 to 7.9]
  Hospitalizations/ER Annualized rate (total) | 2.46 [0.0 to 22.1] | 1.44 [0.0 to 7.9]
  Hospitalizations/ER Annualized rate (VOC related) | 2.27 [0.0 to 22.1] | 0.48 [0.0 to 7.9]

8. Secondary Outcome: Annualized Days of Total and VOC-related Hospitalizations and Emergency Room (ER) Visits
Description: Assess the efficacy of crizanlizumab at 5.0 mg/kg and 7.5 mg/kg in SCD patients for hospitalizations and ER visits. Annualized days of all hospitalizations and ER visits = Number of days of all hospitalizations and ER visits × 365.25/(End date - treatment start date + 1).
  End date is defined as the minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-glutamine or other therapies such as voxelotor and to treat SCD and or to prevent/reduce VOCs, cut-off date).
Time Frame: Baseline (Week 1) through approx. 45 months (median exposure to treatment)
Population: as for outcome 5
Measure: Median (Full Range); unit: number of days per year
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg
Number analyzed (Participants) | 45 | 12
number of days per year
  Annualized days (total) | 11.95 [0.0 to 86.2] | 3.17 [0.0 to 36.8]
  Annualized days (VOC related) | 9.03 [0.0 to 86.2] | 1.57 [0.0 to 36.8]
  Hospitalizations/ER Annualized days (total) | 10.31 [0.0 to 69.4] | 2.57 [0.0 to 36.8]
  Hospitalizations/ER Annualized days (VOC related) | 7.27 [0.0 to 69.4] | 0.60 [0.0 to 36.8]

9. Secondary Outcome: Annualized Rate of Each Subcategory of All VOC Events (Acute Chest Syndrome (ACS), Priapism, Uncomplicated Sickle Cell-vaso-occlusive Cisis (Uncomplicated SC-VOCs))
Description: Assess the efficacy of crizanlizumab at 5.0 mg/kg and 7.5 mg/kg in SCD patients. The baseline (BL) annualized rate of VOC is defined as the number of VOCs reported in the last 12 months in the eCRF. Annualized rate of VOC=(Number of VOC reported until End date ×365.25)/(End date - date of first dose of study treatment+1).
  End date is defined as the minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-glutamine or other therapies such as voxelotor and erythropoietin to treat SCD and or to prevent/reduce VOCs, cut-off date).
Time Frame: Baseline (Week 1) through approx. 45 months (median exposure to treatment)
Population: as for outcome 5
Measure: Median (Full Range); unit: number of events per year
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg
Number analyzed (Participants) | 45 | 12
number of events per year
  BL annualized rate of VOC: ACS: number analyzed (Participants) | 11 | 5
  BL annualized rate of VOC: ACS | 0.00 [0.0 to 2.0] | 0.00 [0.0 to 2.0]
  Annualized rate of VOC on treatment: ACS: number analyzed (Participants) | 11 | 5
  Annualized rate of VOC on treatment: ACS | 0.62 [0.0 to 2.7] | 0.25 [0.0 to 0.6]
  BL annualized rate of VOC: Priapism: number analyzed (Participants) | 3 | 0
  BL annualized rate of VOC: Priapism | 1.00 [0.0 to 4.0] |
  Annualized rate of VOC on treatment: Priapism: number analyzed (Participants) | 3 | 0
  Annualized rate of VOC on treatment: Priapism | 1.58 [0.0 to 3.8] |
  BL annualized rate of VOC: Uncomplicated SC-VOCs: number analyzed (Participants) | 44 | 11
  BL annualized rate of VOC: Uncomplicated SC-VOCs | 3.00 [1.0 to 25.0] | 2.00 [1.0 to 9.0]
  Annualized rate of VOC on treatment: Uncomplicated SC-VOCs: number analyzed (Participants) | 44 | 11
  Annualized rate of VOC on treatment: Uncomplicated SC-VOCs | 2.58 [0.0 to 17.3] | 1.04 [0.0 to 7.9]

10. Secondary Outcome: Annualized Rate of VOC Events (Including Both Healthcare Visit and Home Treatment)
Description: Assess the efficacy of crizanlizumab at 5.0 mg/kg and 7.5 mg/kg in SCD patients. Annualized rate of VOC=(Number of VOC reported until End date ×365.25)/(End date -date of first dose of study treatment+1).
  End date is defined as th e minimum of (last dose date until treatment discontinuation + 27 days, date of initiation or discontinuation of HU/HC or L-glutamine or other therapies such as voxelotor and erythropoietin to treat SCD and or to prevent/reduce VOCs, cut-off date).
Time Frame: Baseline (Week 1) through approx. 45 months (median exposure to treatment)
Population: as for outcome 5
Measure: Median (Full Range); unit: number of events per year
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg
Number analyzed (Participants) | 45 | 12
number of events per year | 3.42 [0.0 to 17.3] | 1.65 [0.0 to 9.3]

11. Secondary Outcome: Number of Participants With Immunogenicity (IG) by Any Positive Status
Description: Assess safety and tolerability of crizanlizumab at 5.0 mg/kg and 7.5 mg/kg in SCD patients by the percentage of participants with any positive status. Immunogenicity is the measurement of anti-drug antibodies (ADA) to crizanlizumab.
Time Frame: Baseline (Week 1), post-baseline (approx. 45 months (median exposure))
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- All Participants: Participants were administered either crizanlizumab at a dose of 5.0 mg/kg or at 7.5 mg/kg by IV infusion.
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg | All Participants
Number analyzed (Participants) | 45 | 12 | 57
Participants
  Baseline: Positive | 0 | 0 | 0
  Post-Baseline: Any Positive | 0 | 0 | 0

12. Primary Outcome: Percentage of P-selectin Inhibition Prior to Each Study Drug Dose of Crizanlizumab at 5.0 mg/kg in Sickle Cell Disease (SCD) Patients
Description: To characterize the PD effect of crizanlizumab in terms of Percentage of P-selectin inhibition prior to study drug dose at 5 mg/kg in CSD patients.
Time Frame: Pre-dose on Day 1 for Weeks 3, 7, 11, 15, 19, 23, 27, 31,35, 39, 43, 47, 51 (at 0 hr or pre-dose)
Population: Patients in the PD analysis set 2 (PDS2) with an available value for the outcome measure. PDS2 included all patients who received at least one planned treatment of 5.0 mg/kg and provided at least one corresponding evaluable PD assessment.
Measure: Mean (Standard Deviation); unit: percentage of P-selectin inhibition
Arm/Group | Crizanlizumab 5.0 mg/kg
Number analyzed (Participants) | 44
percentage of P-selectin inhibition
  Week (W) 3 Day (D) 1: 0 hrs pre-dose: number analyzed (Participants) | 38
  Week (W) 3 Day (D) 1: 0 hrs pre-dose | 97.3 (7.49)
  W7D1: 0 hrs pre-dose: number analyzed (Participants) | 41
  W7D1: 0 hrs pre-dose | 93.0 (17.1)
  W11D1: 0 hrs pre-dose: number analyzed (Participants) | 40
  W11D1: 0 hrs pre-dose | 87.8 (22.6)
  W15D1: 0 hrs pre-dose: number analyzed (Participants) | 37
  W15D1: 0 hrs pre-dose | 94.1 (12.8)
  WD19: 0 hrs pre-dose: number analyzed (Participants) | 35
  WD19: 0 hrs pre-dose | 91.7 (18.5)
  W23D1: 0 hrs pre-dose: number analyzed (Participants) | 37
  W23D1: 0 hrs pre-dose | 93.2 (14.9)
  W27D1: 0 hrs pre-dose: number analyzed (Participants) | 35
  W27D1: 0 hrs pre-dose | 94.3 (13.0)
  W31D1: 0 hrs pre-dose: number analyzed (Participants) | 35
  W31D1: 0 hrs pre-dose | 92.4 (18.9)
  W35D1: 0 hrs pre-dose: number analyzed (Participants) | 32
  W35D1: 0 hrs pre-dose | 91.7 (14.7)
  W39D1: 0 hrs pre-dose: number analyzed (Participants) | 34
  W39D1: 0 hrs pre-dose | 88.5 (21.2)
  W43D1: 0 hrs pre-dose: number analyzed (Participants) | 34
  W43D1: 0 hrs pre-dose | 86.1 (24.8)
  W47D1: 0 hrs pre-dose: number analyzed (Participants) | 34
  W47D1: 0 hrs pre-dose | 92.1 (16.8)
  W51D1: 0 hrs pre-dose: number analyzed (Participants) | 33
  W51D1: 0 hrs pre-dose | 91.5 (17.6)

ADVERSE EVENTS:
Time Frame: All deaths, Serious Adverse Events, and Other Adverse Events for both 'Treatment phase' and 'Post-treatment follow-up phase' (up to 105 days after the last dose of study treatment) were reported. The median duration of exposure to crizanlizumab was 206.1 weeks in the 5.0 mg/kg dose group and 169.6 weeks in the 7.5 mg/kg dose group.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up.
  Other Adverse Event: An adverse event that is not a serious adverse event, meaning that it does not result in death, is not life-threatening, does not require inpatient hospitalization or extend a current hospital stay, does not result in an ongoing or significant incapacity or interfere substantially with normal life functions, and does not cause a congenital anomaly or birth defect.
Arm/Group | Crizanlizumab 5.0 mg/kg | Crizanlizumab 7.5 mg/kg | All Participants
All-Cause Mortality (participants affected / at risk) | 1/45 | 1/12 | 2/57
Serious Adverse Events (participants affected / at risk) | 22/45 | 6/12 | 28/57
Other Adverse Events (participants affected / at risk) | 42/45 | 11/12 | 53/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab 5.0 mg/kg (N=45) | Crizanlizumab 7.5 mg/kg (N=12) | All Participants (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Cytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1
Tooth erosion (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 2
Gait disturbance (General disorders) | 1 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 1
Arthritis infective (Infections and infestations) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 3 | 1 | 4
Cystitis (Infections and infestations) | 1 | 0 | 1
Device related bacteraemia (Infections and infestations) | 1 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0 | 3
Rhinovirus infection (Infections and infestations) | 1 | 0 | 1
Salmonella bacteraemia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 2
Wound sepsis (Infections and infestations) | 1 | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizanlizumab 5.0 mg/kg (N=45) | Crizanlizumab 7.5 mg/kg (N=12) | All Participants (N=57)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 2
Tornwaldt cyst (Congenital, familial and genetic disorders) | 0 | 1 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 2 | 1 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 1
Retinal drusen (Eye disorders) | 0 | 1 | 1
Retinopathy sickle cell (Eye disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 3
Constipation (Gastrointestinal disorders) | 3 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 6
Gastritis (Gastrointestinal disorders) | 3 | 0 | 3
Nausea (Gastrointestinal disorders) | 6 | 2 | 8
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 4 | 0 | 4
Vomiting (Gastrointestinal disorders) | 4 | 3 | 7
Chest pain (General disorders) | 6 | 1 | 7
Drug withdrawal syndrome (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 4 | 1 | 5
Oedema peripheral (General disorders) | 6 | 0 | 6
Pain (General disorders) | 2 | 1 | 3
Peripheral swelling (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 13 | 3 | 16
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1
Ocular icterus (Hepatobiliary disorders) | 1 | 2 | 3
Acute sinusitis (Infections and infestations) | 2 | 1 | 3
COVID-19 (Infections and infestations) | 5 | 2 | 7
Cystitis (Infections and infestations) | 2 | 1 | 3
Gastroenteritis (Infections and infestations) | 3 | 1 | 4
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2
Otitis media acute (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 4 | 1 | 5
Pneumonia (Infections and infestations) | 2 | 1 | 3
Tooth infection (Infections and infestations) | 3 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 10 | 2 | 12
Urinary tract infection (Infections and infestations) | 4 | 0 | 4
Post-traumatic pain (Injury, poisoning and procedural complications) | 3 | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 5 | 2 | 7
Skin laceration (Injury, poisoning and procedural complications) | 2 | 1 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 3
Haematocrit decreased (Investigations) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 4
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 2 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 2 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 7
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0 | 6
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Headache (Nervous system disorders) | 12 | 2 | 14
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 2 | 2 | 4
Depression (Psychiatric disorders) | 2 | 1 | 3
Insomnia (Psychiatric disorders) | 4 | 0 | 4
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2
Dysuria (Renal and urinary disorders) | 3 | 0 | 3
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Hypertension (Vascular disorders) | 4 | 0 | 4

LIMITATIONS AND CAVEATS:
This study provided a 5-year follow up (f/u) data that fully characterized the safety, tolerability & treatment of the 5.0 mg/kg & 7.5 mg/kg doses of crizanlizumab along with the initially planned PK & PD data. As the goal of study f/u was reached, study was considered completed & it was in line with the end of study as defined in the study protocol, the sponsor closed the study as the participants were no longer receiving intervention or being examined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03264989/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT03264989/SAP_000.pdf